CLINICAL TRIAL: NCT00978406
Title: National Cancer Institute (NCI) Food Study
Brief Title: National Cancer Institute Food Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909209; 09-C-N209
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Validation Study; Diet Surveys; Nutritional Assessment; Epidemiology; Methodologic Study
Keywords: Dietary Assessment Methods; Measurement of Diet; 24-Hour Diet Recall; Validation; Feeding Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy volunteers

SUMMARY:
Information about Americans food choices and opinions helps researchers and law makers to develop policies and programs to promote health. For this reason, it is important to be able to collect good quality information about how people think about food. This project will compare different ways of collecting information about food from adults.

DETAILED DESCRIPTION:
Objectives:

-To compare different ways of collecting information about food choices and opinions from adults.

Eligibility:

* Individuals between the ages of 20 and 70, recruited from a database of volunteers who wish to participate in research studies.
* Volunteers must have high-speed Internet access.
* Individuals who have previously been involved in a research study will be excluded.

Design:

-Participants will come to a research study center for three consecutive meals (approximately 45 minutes per meal). On the following day, participants will return to the study center for an interview about their food choices and opinions (approximately 45 minutes).

ELIGIBILITY:
* Eligibility Criteria
* Individuals between the ages of 20 and 70, recruited from a database of volunteers who wish to participate in research studies.
* Volunteers must have high-speed Internet access.
* Individuals who have previously been involved in a research study will be excluded.
* Subjects will be accrued from a variety of racial and ethnic groups and of varying educational achievement, though these characteristics will not be used to assess eligibility.
* All subjects will provide informed consent.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers living in Maryland@@@
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2009-08-26 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Agreement of truth and reported dietary intake | 2 days
  Measured exact intake of foods will be compared to reported intake by the participant. Two different reporting systems will be compared with truth.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Potischman, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Westat, Inc., Rockville, Maryland, United States

REFERENCES:
- [Derived] Kirkpatrick SI, Potischman N, Dodd KW, Douglass D, Zimmerman TP, Kahle LL, Thompson FE, George SM, Subar AF. The Use of Digital Images in 24-Hour Recalls May Lead to Less Misestimation of Portion Size Compared with Traditional Interviewer-Administered Recalls. J Nutr. 2016 Dec;146(12):2567-2573. doi: 10.3945/jn.116.237271. Epub 2016 Nov 2. PMID 27807039
- [Derived] Kirkpatrick SI, Subar AF, Douglass D, Zimmerman TP, Thompson FE, Kahle LL, George SM, Dodd KW, Potischman N. Performance of the Automated Self-Administered 24-hour Recall relative to a measure of true intakes and to an interviewer-administered 24-h recall. Am J Clin Nutr. 2014 Jul;100(1):233-40. doi: 10.3945/ajcn.114.083238. Epub 2014 Apr 30. PMID 24787491